CLINICAL TRIAL: NCT04109170
Title: Dry Eye Evaluation System Based on Bioinformatics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huaxia Eye Hospital Group (Other)
Responsible Party: Sponsor
Other Study IDs: FSHX2019-01
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Dry Eye
Keywords: Dry Eye; Bioinformatics; Data mining
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dry Eye Group: This group of subjects were diagnosed with dry eye.
- Normal Control Group: This group of subjects had no dry eye symptoms and signs and belonged to the normal control group.

SUMMARY:
Dry eye is a common ocular surface disease of multifactorial etiology characterized by elevated tear osmolality and inflammation leading to a disrupted ocular surface. The latter is a risk factor for ocular surface infection, yet overt infection is not commonly seen clinically in the typical dry eye patient. This suggests that important innate mechanisms operate to protect the dry eye from invading pathogens. Understand the pathogenesis of dry eye will be the measure to prevention and treatment of dry eye.

In this essay, the investigators use the data of experiment in the patients with dry eye and normal, acquire their tear production, tear film stability, and surface damage. The investigators use weka to calculate the prediction accuracy of the 6 algorithm and select the best one, optimize the parameters to get the final prediction accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Dye Eye

Exclusion Criteria:

* systemic disease (such as diabetes, glaucoma, or systemic collagen vascular disease), ocular disease, a history of tear supplement usage or contact lens wear during the past year,and pregnancy

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People who meet the experimental conditions among the outpatients in our hospital will be selected into the group
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2019-12-23 (Estimated); Study Completion 2020-01-23 (Estimated)

PRIMARY OUTCOMES:
OSDI | up to 2 months
  The Ocular Surface Disease Index (OSDI; Allergan Inc., Irvine, CA)consists of a 12-item questionnaire and is used to assess dry eye disease; the OSDI questions are drawn from three different categories: vision-related functions, ocular symptoms and environmental triggers. The OSDI is scored on a 4-point scale from 0 (indicating no problems) to 4 (indicating a significant problem). Responses to all of the questions are combined to generate a composite OSDI score that ranges from 0 to 100, with higher OSDI scores representing greater disability. Subjects were asked questions regarding the dry eye symptoms that they experience.
Schirmer I test | up to 2 months
  The Schirmer I test (SIT) without anesthesia for tear secretion function was conducted by placing a 30-mm sterile Schirmer Tear Test strip into the junction of the middle and lateral thirds of the inferior fornix of each eye for 5 minutes. The wet portion of the strip was subsequently measured, with lower scores indicating less tear production.
Fluorescein staining | up to 2 months
  The cornea was divided into upper, lower, nasal, temporal and central zones. Superficial punctate keratopathy (SPK) in the cornea was scored from 0 to 3 in each area. Where 0 indicated no staining in the cornea; 1,<5 punctate stains; 2,5-10 punctate stains; and 3,>10 or filamentous staining detected. The total score was recorded by adding the scores of the five zones for each eye (range: 0-15).
Noninvasive Tear Breakup Time | up to 2 months
  Noninvasive Tear Breakup Time (NI-TBUT) measurements of subjects' eyes were obtained by Keratograph 5. At the start of the recording, the patients were asked to blink three times and then keep their eyes open as long as possible. Irregularities in the reflected image indicated the instability of the tear film. Meanwhile, the examination was recorded on video and a single eye of each subject was assessed three times. All the tests were performeded the same temperature and humidity conditions.

SECONDARY OUTCOMES:
Tear meniscus height | up to 2 months
  Tear meniscus height was also performed by the Keratograph 5 and the image of tear meniscus height was obtained by the instrument. The observer measured the tear meniscus height the center of the lower lid margin. This evaluation was taken three times and the average value was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Zhang, PhD,MD, Principal Investigator — Huaxia Eye Hospital of Foshan
Locations (1):
- Huaxia Eye Hosptial of Foshan, Foshan, Guangdong, China